CLINICAL TRIAL: NCT02501148
Title: A Multi-Center Study to Evaluate Acute Safety and Clinical Performance of Paladin® Carotid Post-Dilation Balloon System With Integrated Embolic Protection
Status: Completed | Type: Observational
Sponsor: Contego Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP-1001
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Carotid Artery Stenoses
Keywords: Embolic protection; Carotid artery stenting
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carotid artery stenting: Symptomatic and asymptomatic subjects requiring carotid artery stenting, post-dilation performed using the Paladin System with integrated embolic protection
  Interventions: Device: carotid artery stenting

INTERVENTIONS:
Device: carotid artery stenting — Post-dilation of deployed self-expanding carotid stent with the Paladin Post-Dilation Balloon System with Integrated Embolic Protection
  Other Names: Paladin Post-Dilation Balloon System with Integrated Embolic Protection

SUMMARY:
The purpose of this study is to assess the safety and clinical performance of Paladin System in patients with carotid artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Documented stenotic atherosclerotic lesion located at carotid bifurcation and / or proximal internal carotid artery (ICA)
* Subject is either (A) symptomatic within 6 months of procedure, with an ipsilateral carotid stenosis ≥ 50% by angiography, or (B) asymptomatic with carotid stenosis ≥ 70% by angiography
* Target lesion can be covered by a single stent of no more than 40 mm in length
* Target lesion reference vessel diameter (RVD) is 4.0 mm - 7.0mm
* Sufficient landing zone required for successful deployment of integrated embolic protection filter
* Willing to comply with all follow-up required study visits
* Provision of written informed consent before index procedure

Exclusion Criteria:

* Life expectancy of less than one year
* An evolving, acute or recent stroke within 14 days of study evaluation
* Acute myocardial infarction within 72 hours before procedure
* Known sensitivity to contrast media that cannot be adequately controlled with pre-medication
* Subject has a total occlusion of target carotid artery
* Subject has a previously place stent in ipsilateral carotid artery
* Severe circumferential lesion calcification that may restrict full deployment of carotid stent
* Presence of filling defect or thrombus in target vessel
* Presence of "string sign" of target vessel
* Carotid (intracranial) stenosis located distal to target lesion
* Greater than 50% stenosis of common carotid artery proximal to target lesion.
* Known mobile plaque in aortic arch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults; either gender; requiring percutaneous intervention of an asymptomatic (> 70%) or symptomatic (>50%) internal carotid artery stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Device-related MAE | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Thomas Zeller, MD, Principal Investigator — Universitäts Herzzentrum Freiburg Bad-Krozingen; Prof. Horst Sievert, MD, Principal Investigator — CardioVascular Center, Sankt Katharinen Hospital
Locations (5):
- Germany (5):
  - Universitäts-Herzzentrum Bad Krozingen, Bad Krozingen
  - Sankt Gertrauden Krankenhaus, Berlin
  - CardioVascular Centre Frankfurt, Frankfurt
  - Medizinisches Versorgungszentrum Prof. Mathey, Prof. Schofer GmbH, Hamburg
  - Universitätsklinikum Leipzig, Leipzig

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langhoff R, Schofer J, Scheinert D, Schmidt A, Sedgewick G, Saylors E, Sachar R, Sievert H, Zeller T. Double Filtration During Carotid Artery Stenting Using a Novel Post-Dilation Balloon With Integrated Embolic Protection. JACC Cardiovasc Interv. 2019 Feb 25;12(4):395-403. doi: 10.1016/j.jcin.2018.11.039. PMID 30784647
- See also: Double Filtration During Carotid Artery Stenting Using a Novel Post-Dilation Balloon With Integrated Embolic Protection — https://doi.org/10.1016/j.jcin.2018.11.039